CLINICAL TRIAL: NCT00704470
Title: Excellence in Performance and Stress Reduction During Two Different Full Scale Simulator Training Courses: A Pilot Study
Brief Title: Performance and Stress During Full Scale Simulator Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Dr. Michael Mueller, Dept. of Anesthesiology, University of Technology, Dresden
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: EK261122004
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Performance in Simulated Emergencies; Stress During Simulator Scenario; Behaviour of Physicians in Simulated Emergencies
Keywords: Patient Simulation; Education, Medical, Continuing; Education, Medical, Graduate; Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Classic one-day simulator training for intensivists.
  Interventions: Other: Medical simulator training
- 2 (Experimental): Crew resource management training
  Interventions: Other: Simulator based crew resource management course

INTERVENTIONS:
Other: Medical simulator training — Contains seminars on airway management, general anesthesia, peri-arrest arrhythmias, and advanced life support. Furthermore, participants train in simulator scenarios. In the debriefing instructors discuss management of the critical incidents using videotapes of the scenarios.
  Arms: 1
Other: Simulator based crew resource management course — Contains seminars on human error and non-technical skills. Furthermore, participants train in simulator scenarios. In the debriefing instructors discuss usage of non-technical skills as well as behaviour of the participants using videotapes of the scenarios.
  Arms: 2

SUMMARY:
In Intensive Care Medicine, critical incidents are not rare and may result in fatal outcome. High fidelity patient simulators are commonly used in training curricula for healthcare professionals especially in anesthesiology, emergency medicine, and intensive care medicine. Several different course concepts have previously been published. As we know from recently published data, up to 80% of all critical incidents in the field of medicine are caused by human error. The authors of the present study aimed to investigate the effects of two different course concepts (one addressing technical skills in intensive care medicine and on addressing non-technical skills) on stress and performance. Stress and performance are measured in a pre-intervention and a post-intervention testing scenario.

ELIGIBILITY:
Inclusion Criteria:

* Physician with experience in intensive care medicine.

Exclusion Criteria:

* No experience in intensive care medicine
* previously taken part in simulator training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Performance in simulated emergencies (medical performance and non-technical skills)

SECONDARY OUTCOMES:
Stress in simulated emergencies (measured by salivary amylase and cortisol levels)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Mueller, MD, Principal Investigator — Director of Simulation Centre, Dept. of Anesthesiology, University Hospital Dresden
Locations (1):
- Interdisciplinary Medical Simulation Centre, University Hospital Dresden, Dresden, Germany

REFERENCES:
- [Background] Muller MP, Hansel M, Stehr SN, Fichtner A, Weber S, Hardt F, Bergmann B, Koch T. Six steps from head to hand: a simulator based transfer oriented psychological training to improve patient safety. Resuscitation. 2007 Apr;73(1):137-43. doi: 10.1016/j.resuscitation.2006.08.011. Epub 2007 Jan 22. PMID 17241735
- See also: Website of Interdisciplinary Medical Simulation Centre — http://www.isimed.info